CLINICAL TRIAL: NCT02482987
Title: Comparison of Two Different Alveolar Ridge Preservation Techniques
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Eisenhower Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Brandon Coleman, Assistant Director, Advanced Education Program in Periodontics, Eisenhower Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 408953-1
Record Dates: First submitted 2015-06-19; First posted 2015-06-26 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Loss of Teeth Due to Extraction
Keywords: dental; extraction; socket preservation; ridge preservation; implant site preparation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cytoplast (Experimental): Patients will receive ridge preservation procedure with a Cytoplast barrier membrane
  Interventions: Device: dense polytetrafluoroethylene (dPTFE) membrane Cytoplast; Procedure: Ridge Preservation with overlay graft; Procedure: Ridge Preservation without overlay graft
- BioXclude (Experimental): Patients will receive ridge preservation procedure with a BioXclude barrier membrane
  Interventions: Device: human amniotic-tissue derived membrane BioXclude; Procedure: Ridge Preservation with overlay graft; Procedure: Ridge Preservation without overlay graft

INTERVENTIONS:
Device: dense polytetrafluoroethylene (dPTFE) membrane Cytoplast — ridge preservation intervention using the dPTFE membrane device
  Other Names: Cytoplast
  Arms: Cytoplast
Device: human amniotic-tissue derived membrane BioXclude — ridge preservation intervention using the dPTFE membrane device
  Other Names: BioXclude
  Arms: BioXclude
Procedure: Ridge Preservation with overlay graft — ridge preservation intervention with additional freeze dried bone allograft (FDBA) placed buccal to the socket
Procedure: Ridge Preservation without overlay graft — ridge preservation without overlay graft / traditional FDBA placement into the socket only

SUMMARY:
The purpose of this study is to compare two barrier membrane products, Cytoplast (dPTFE) and BioXclude (human amnion chorion allograft), for their relative efficacies in dental socket preservation procedures, both when the socket is filled and overfilled with freeze dried bone allograft (FDBA).

DETAILED DESCRIPTION:
This single-blind, randomized clinical trial aims to compare two different, commercially available materials to assess their relative efficacies in socket preservation procedures after tooth extraction. Patients presenting with single teeth deemed clinically hopeless and treatment planned for removal in the normal course of clinical dentistry will be considered for this study. If eligible, a ridge/socket preservation procedure will be performed at the time of extraction. Periodontics residents will perform the procedure under the supervision of board certified staff. Patients will be randomized via concealed random number sequence into one of four groups, based on a combination of materials and graft placement techniques. Patients will be equally distributed into the following groups: (1) dense polytetrafluoroethylene (Cytoplast) (2) Cytoplast with additional buccal augmentation/onlay graft, (3) human amniotic-tissue derived membrane (BioXclude), and (4) BioXclude with additional buccal augmentation/onlay graft. All four treatment groups are consistent with the current standard of care, and this study seeks to compare techniques and materials as part of routine, clinical/periodontal therapy in order to determine superiority. Approximately 150 patients will be enrolled and distributed equally among the four groups. Any post-operative complications will be managed and documented during follow-up appointments at 1, 2 and 4 weeks. Cone beam computed tomography (CBCT) will be used as the primary assessment tool, and scans will be compared between a pre-operative baseline time point and a scan taken after 4 months of healing to prepare for implant placement. The primary dependent variables will be (1) percent of baseline alveolar ridge changes (both horizontal and vertical) and (2) whether or not the anticipated dental implant could be placed appropriately. Secondary outcomes include ease of use, perceptions of pain, complications, cost-effectiveness, and changes in keratinized tissue.

ELIGIBILITY:
Inclusion Criteria:

* All active duty military patients (age 18-65) referred to the investigators' facility's periodontics department for diagnosis of "hopeless" tooth with documented confirmation of diagnosis by periodontal staff
* Eligible for extraction and ridge preservation (adequately healthy and not otherwise disqualified)

Exclusion Criteria:

* Pregnant or breastfeeding
* History of allergy to involved products
* Current acute infection at the site (chronic periapical infections will not exclude the patient)
* Elian Type 3 extraction sockets
* Sites not treatment planned for implant therapy
* Third molar sites
* American Society of Anesthesiology Category III patients (medically compromised)
* Active duty military patients in a student status

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-07; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Alveolar Ridge Width | from baseline to final cone beam CT scan (approximately 4 months)
  Alveolar ridge dimensional change (horizontal) from Cone beam CT
Alveolar Ridge Height | from baseline to final cone beam CT scan (approximately 4 months)
  Alveolar ridge dimensional change (vertical) from cone beam CT

SECONDARY OUTCOMES:
Post-operative pain perception | 1 week after surgical extraction procedure
  self-report by patient on visual analog scale
Platform size of implant placed | Implant surgery, approximtely 4 months after baseline
  Whether or not the originally intended implant size could be placed
Keratinized tissue width (baseline) | pre-op / baseline assessment (after randomization)(prior to time=0)
Keratinized tissue width (final) | from pre-op assessment at time of randomization to implant surgery (4 months)
Elian classification (anticipated) | pre-op / baseline assessment (after randomization)(prior to time=0)
  Operators will report an anticipated socket preservation classification according to Elian 2007
Elian classification (actual) | intra-operative surgical finding (extraction surgery)(time=0)
  Operators will report the actual socket preservation classification according to Elian 2007
Buccal plate thickness | intra-operative surgical finding (extraction surgery)(time = 0)
  intra-operative measurements, presence or absence of a dehiscence / fenestration
Buccal plate fenestration | intra-operative surgical finding (extraction surgery)(time = 0)
  determined at time of extraction surgery, and noted as a possible confounding variable
Complications after surgery (infection) | 0-4 months
  infection, determined by presence of purulence, lymphadenopathy and/or febrile status
Complications after surgery (membrane exfoliation) | 0-4 months
  dichotomous variable, presence or absence of the membrane for the duration of the study
Peri-operative clinician's report (extraction difficulty) | intra-operative surgical finding (extraction surgery)
  subjective extraction difficulty, as reported by the clinician

OTHER OUTCOMES:
Sedation utilization | intra-operative surgical variable (determined in advance, at baseline)
  presence or absence of sedation drugs during the procedure
Cost | 0-4 months
  cost/benefit for each product

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Coleman, DDS,MS, Principal Investigator — US Army Fort Gordon DENTAC
Locations (1):
- Tingay Dental Clinic, Fort Gordon, Georgia, United States